CLINICAL TRIAL: NCT01817075
Title: Impact of Cleansing With Chlorhexidine Gluconate (CHG) on Reducing Central Line Associated Bloodstream Infection (CLABSI) and Acquisition of Multi-drug Resistant Organisms (MDRO) in Children With Cancer or Those Receiving Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Chlorhexidine Gluconate Cleansing in Preventing Central Line Associated Bloodstream Infection and Acquisition of Multi-drug Resistant Organisms in Younger Patients With Cancer or Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCL1034; NCI-2013-00595 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL1034 (Other: Childrens Oncology Group); COG-ACCL1034 (Other: DCP); ACCL1034 (Other: CTEP); R01CA163394 (NIH); U10CA095861 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2020-03

CONDITIONS: Bacterial Infection; Benign Neoplasm; Malignant Neoplasm; Methicillin-Resistant Staphylococcus Aureus Infection; Myeloid Neoplasm; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Bacterial Infections; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (CHG cleansing wipe) (Experimental): Patients receive CHG cleansing with topical skin wipes QD for 90 days.
  Interventions: Procedure: Chlorhexidine Gluconate Skin Cleanser; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm II (control) (Active Comparator): Patients receive control cleansing with topical skin wipes QD for 90 days.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Mild Soap Skin Cleanser; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Chlorhexidine Gluconate Skin Cleanser — Given CHG cleansing
  Other Names: Skin Cleanser with Chlorhexidine Gluconate
  Arms: Arm I (CHG cleansing wipe)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Mild Soap Skin Cleanser — Given control cleansing
  Other Names: Skin Cleanser with Mild Soap
  Arms: Arm II (control)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies chlorhexidine gluconate cleansing to see how well it works compared to control cleansing in preventing central line associated bloodstream infection and acquisition of multi-drug resistant organisms in younger patients with cancer or undergoing donor stem cell transplant. Chlorhexidine gluconate may help reduce bloodstream infections and bacterial infections associated with the central line.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether chlorhexidine gluconate (CHG) cleansing decreases central line associated bloodstream infection (CLABSI) in children with cancer or those receiving an allogeneic hematopoietic cell transplantation (HCT).

SECONDARY OBJECTIVES:

I. To determine whether CHG cleansing decreases acquisition of multi-drug resistant organisms (MDRO: vancomycin resistant enterococci [VRE], methicillin resistant Staphylococcus aureus [MRSA], etc.) in children with cancer or those receiving allogeneic HCT.

II. To determine whether CHG cleansing in children with cancer or those receiving allogeneic HCT is associated with cutaneous bacterial isolates with reduced susceptibility to CHG.

III. To determine whether CHG cleansing decreases positive blood cultures in children with cancer or those receiving allogeneic HCT.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive CHG cleansing with topical skin wipes once daily (QD) for 90 days.

ARM II: Patients receive control cleansing with topical skin wipes QD for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* TRANSPLANT PATIENTS: all patients undergoing planned allogeneic transplant (both malignant and non-malignant diagnoses)
* ONCOLOGY PATIENTS: patients with an oncology diagnosis that are or will be on a chemotherapy regimen that will last for an additional >= 3 months or are on or will be on a chemotherapy regimen for < 3 months and then proceed to transplant (allogeneic or autologous stem cell rescue) during the 3-month study period
* Patients undergoing allogeneic transplant must have, or be scheduled to have, an external tunneled central venous catheter (CVC) (Broviacs, Hickmans, tunneled percutaneously inserted central catheter [PICCs], etc.) and/or non-tunneled percutaneously inserted central catheter (PICC) that is expected to remain in place for an additional >= 3 months
* Patients with acute myelogenous leukemia (AML) or relapsed acute lymphoblastic leukemia (ALL) that will receive chemotherapy with/without transplant must have, or be scheduled to have, an external tunneled CVC (Broviacs, Hickmans, tunneled PICCs, etc.) and/or non-tunneled PICC that is expected to remain in place for an additional >= 3 months
* All other oncology patients that will receive chemotherapy with/without transplant must have, or be scheduled to have, an external tunneled CVC (Broviacs, Hickmans, tunneled PICCs, etc.) that is expected to remain in place for an additional >= 3 months
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with a previous or current line infection are ineligible until 14 days after the completion of antibiotics
* Patients with only totally implanted CVCs or ports are ineligible
* Patients with a known allergy or hypersensitivity to CHG are ineligible
* Patients with chronic, severe, generalized skin breakdown (such as generalized blistering, burns, severe graft versus host disease [GVHD] with open sores, etc.) are ineligible
* Patients currently enrolled on Children's Oncology Group (COG) study ACCL0934 are not eligible until they have completed the infection observation period of that study
* Patients scheduled to receive broad-spectrum prophylactic antibacterial therapy are ineligible; patients only receiving prophylaxis for Pneumocystis pneumonia (PCP) (trimethoprim [TMP]/sulfamethoxazole [SMX]) or encapsulated organisms (penicillin) are eligible
* Patients receiving sorafenib at the time of enrollment and those who are scheduled to receive sorafenib as part of a treatment plan are ineligible
* Patients using prophylactic antimicrobial locks in the CVC at the time of enrollment and those who are scheduled to receive antimicrobial locks in the CVC as part of a treatment plan are ineligible
* Patients previously enrolled on this trial are ineligible
* Females who are pregnant or breastfeeding are ineligible

Ages: 2 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Zerr, Principal Investigator — Children's Oncology Group
Locations (59):
- United States (53):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
- Canada (4):
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (CHG Cleansing Wipe) | Arm II (Control)
Started | 88 | 89
Completed | 41 | 54
Not Completed | 47 | 35
Not completed — Adverse Event | 7 | 5
Not completed — Physician Decision | 9 | 12
Not completed — Withdrawal by Subject | 31 | 15
Not completed — Received Sorafenib after enrollment | 0 | 1
Not completed — Ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (CHG Cleansing Wipe) | Arm II (Control) | Total
Number analyzed (Participants) | 88 | 89 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 83 | 88 | 171
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.4 (5.8) | 5 (4.8) | 6.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 53 | 53 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 20 | 36
  Not Hispanic or Latino | 69 | 63 | 132
  Unknown or Not Reported | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 14 | 9 | 23
  White | 51 | 54 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 21 | 36
Region of Enrollment [Number; unit: participants]
  United States | 77 | 82 | 159
  Canada | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Central Line-associated Bloodstream Infections (CLABSI) Events During the At-risk Days
Description: Rate of CLABSI per 1000 at-risk days. CLABSI outcome is defined according to the January 2015 Centers for Disease Control and Prevention (CDC) criteria. At risk days are defined as days with eligible central lines in place.
Time Frame: Up to 90 days post enrollment date
Population: 3 patients were excluded (2 ineligible and 1 withdrew consent) leaving 174 patients in the analyses.
Measure: Number (95% Confidence Interval); unit: CLABSI per 1000 at-risk days.
Arm/Group | Arm I (CHG Cleansing Wipe) | Arm II (Control)
Number analyzed (Participants) | 88 | 86
CLABSI per 1000 at-risk days. | 5.44 [3.62 to 8.18] | 3.1 [1.82 to 5.28]

2. Secondary Outcome: Percentage of Patients With Multi-drug Resistant Organisms (MDRO)
Description: MDROs are defined as Staphylococcus aureus resistant to oxacillin, Enterococcus spp. resistant to vancomycin, Klebsiella pneumoniae or Escherichia coli non-susceptible (intermediate or resistant) to ceftriaxone, ceftazidime, cefepime or any carbapenem, and Pseudomonas aeruginosa or Acinetobacter baumannii resistant to any carbapenem or ceftazidime, and either an aminoglycoside or fluoroquinolone. Clostridium difficile infection (CDI) is included as an MDRO and is defined as a positive lab test for C. difficile and > 3 unformed stools in < 24 hours.
Time Frame: Up to 90 days post enrollment date
Population: 3 patients were excluded (2 ineligible and 1 withdrew consent) leaving 174 patients in the analyses.
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (CHG Cleansing Wipe) | Arm II (Control)
Number analyzed (Participants) | 88 | 86
Percentage of patients | 15 | 12

3. Secondary Outcome: Percentage of Patients Who Acquire Cutaneous Bacterial Isolates With Reduced Susceptibility to Chlorhexidine Gluconate (CHG)
Description: Susceptibility to CHG is defined by MIC cutoff that is cutaneous staphylococcal isolate isolated from a follow-up swab with CHG MIC > 4 ug/mL in patient without a resistant staphylococcal isolate isolated from a baseline swab.
Time Frame: Up to 90 days post enrollment date
Population: 135 participants contributed a baseline and at least one follow-up swab and were included in this analysis
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (CHG Cleansing Wipe) | Arm II (Control)
Number analyzed (Participants) | 62 | 73
percentage of patients | 17.7 | 5.5

4. Secondary Outcome: Rate of Bacteremia Per 1000 At-risk Days
Description: A bacteremia episode is defined any positive blood culture. At risk days are defined as days with eligible central lines in place.
Time Frame: Up to 90 days post enrollment date
Population: 3 patients were excluded (2 ineligible and 1 withdrew consent) leaving 174 patients in the analysis.
Measure: Number (95% Confidence Interval); unit: bacteremia per 1000 at-risk days
Arm/Group | Arm I (CHG Cleansing Wipe) | Arm II (Control)
Number analyzed (Participants) | 88 | 86
bacteremia per 1000 at-risk days | 7.24 [5.5 to 9.5] | 4.93 [3.5 to 6.9]

ADVERSE EVENTS:
Time Frame: Collected Adverse Events within the 90 day observation period
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible and unevaluable (withdraw of consent) patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm I (CHG Cleansing Wipe) | Arm II (Control)
All-Cause Mortality (participants affected / at risk) | 1/88 | 3/86
Serious Adverse Events (participants affected / at risk) | 0/88 | 2/86
Other Adverse Events (participants affected / at risk) | 22/88 | 14/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (CHG Cleansing Wipe) (N=88) | Arm II (Control) (N=86)
Cardiac arrest (Cardiac disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (CHG Cleansing Wipe) (N=88) | Arm II (Control) (N=86)
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 7
Sepsis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9 | 4
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT01817075/Prot_SAP_000.pdf